CLINICAL TRIAL: NCT03500328
Title: A Pragmatic Trial to Evaluate the Intermediate-term Effects of Early, Aggressive Versus Escalation Therapy in People With Multiple Sclerosis
Brief Title: Traditional Versus Early Aggressive Therapy for Multiple Sclerosis Trial
Acronym: TREAT-MS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00143534
Record Dates: First submitted 2018-02-21; First posted 2018-04-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab; Alemtuzumab; ocrelizumab; Cladribine; ofatumumab; Rituximab; Glatiramer Acetate; Interferons; Injections, Intramuscular; Injections, Subcutaneous; teriflunomide; Fumarates; Fingolimod Hydrochloride; siponimod; ozanimod; ponesimod; Coat Protein Complex I; Interferon beta-1a; Interferon beta-1b; peginterferon beta-1a; Dimethyl Fumarate; diroximel fumarate; monomethyl fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Aggressive Therapy (Active Comparator): Early Aggressive Therapy choices and maximum allowable doses:
  * Natalizumab/natalizumab-sztn (Tysabri/Tyruko), 300 mg IV q 4 wks
  * Alemtuzumab (Lemtrada), 12 mg IV daily (QD) for 5 days; 1 yr later: 12 mg IV QD for 3 days
  * Ocrelizumab (Ocrevus), 300 mg IV every 2 wks (for 2 doses) at initiation; 600 mg IV q 6 mths
  * Rituximab/rituximab biosimilars (Rituxan/Riabni/Truxima/Ruxience), 1000 mg IV every 2 wks (for 2 doses); may repeat q 16-24 wks
  * Cladribine (Mavenclad), 3.5 mg per kg body wt orally divided into 2 yrly tmt courses (1.75 mg per kg body wt each yr); yrly tmt course divided into 2 tmt cycles; administer cycle dose as 1-2 tablets QD over 4-5 days
  * Ofatumumab (Kesimpta), 20 mg SC wkly for wks 0, 1 and 2; 20 mg subcutaneously (SC) mthly starting at wk 4
  * Ublituximab-xiiy (Briumvi), 150 mg IV (1st dose); 450 mg IV 2 wks after first dose; 450 mg IV q 24 wks
  * Ocrelizumab and hyaluronidase-ocsq (Ocrevus Zunovo), 920 mg ocrelizumab and 23,000 U hyaluronidase SC q 6 months
  Interventions: Other: Natalizumab/natalizumab-sztn, Alemtuzumab, Ocrelizumab, Rituximab/rituximab-arrx/rituximab-abbs/rituximab-pvvr, Cladribine, Ofatumumab, Ublituximab-xiiy, Ocrelizumab and hyaluronidase-ocsq
- Traditional Therapy (Active Comparator): Traditional Therapy choices and maximum allowable doses:
  * Glatiramer acetate (Copaxone, Glatopa, and other generics), 20 mg SC daily, or 40 mg SC 3 times a wk
  * Intramuscular (IM) interferon (Avonex), 30 mcg IM weekly
  * SC interferon (Betaseron, Extavia, Rebif), 0.25 mg SC every other day (Betaseron, Extavia); 44 mcg SC 3 times a wk (Rebif)
  * Pegylated interferon (Plegridy), 125 mcg SC every 14 days
  * Teriflunomide (Aubagio), 14 mg PO QD
  * Dimethyl fumarate (Tecfidera and generics), 240 mg PO twice a day (BID)
  * Diroximel fumarate (Vumerity), 462 mg PO BID
  * Monomethyl fumarate (Bafiertam), 190 mg PO BID
  * Fingolimod (Gilenya and generics), 0.5 mg PO QD
  * Siponimod (Mayzent), 1 mg PO QD or 2 mg PO QD
  * Ozanimod (Zeposia), 0.92 mg PO QD
  * Ponesimod (Ponvory), 20 mg PO QD
  * Fingolimod ODT (Tascenso), 0.25 mg PO QD if <=40 kg; 0.5 mg PO QD if > 40 kg
  Interventions: Other: Glatiramer acetate, Interferons (intramuscular, subcutaneous, pegylated) Teriflunomide, Fumarates (dimethyl, diroximel, monomethyl) Fingolimod, Siponimod, Ozanimod, Ponesimod

INTERVENTIONS:
Other: Natalizumab/natalizumab-sztn, Alemtuzumab, Ocrelizumab, Rituximab/rituximab-arrx/rituximab-abbs/rituximab-pvvr, Cladribine, Ofatumumab, Ublituximab-xiiy, Ocrelizumab and hyaluronidase-ocsq — Early Aggressive Therapy
  Other Names: Tysabri, Lemtrada, Ocrevus, Rituxan/Riabni/Truxima/Ruxience, Mavenclad, Kesimpta, Briumvi, Ocrevus Zunovo
  Arms: Early Aggressive Therapy
Other: Glatiramer acetate, Interferons (intramuscular, subcutaneous, pegylated) Teriflunomide, Fumarates (dimethyl, diroximel, monomethyl) Fingolimod, Siponimod, Ozanimod, Ponesimod — Traditional Therapy
  Other Names: Copaxone, Glatopa, Avonex, Betaseron, Extavia, Rebif, Plegridy, Aubagio, Tecfidera, Vumerity, Bafiertam, Gilenya, Mayzent, Zeposia, Ponvory, Tascenso
  Arms: Traditional Therapy

SUMMARY:
FDA-approved multiple sclerosis (MS) disease-modifying therapies (DMTs) target the relapsing phase of MS but have minimal impact once the progressive phase has begun. It is unclear if, in the relapsing phase, there is an advantage of early aggressive therapy with respect to preventing long-term disability. The infectious risks and other complications associated with higher-efficacy treatments highlight the need to quantify their effectiveness in preventing disability.

The TRaditional versus Early Aggressive Therapy for MS (TREAT-MS) trial is a pragmatic, randomized controlled trial that has two primary aims: 1) to evaluate, jointly and independently among patients deemed at higher risk vs. lower risk for disability accumulation, whether an "early aggressive" therapy approach, versus starting with a traditional, first-line therapy, influences the intermediate-term risk of disability, and 2) to evaluate if, among patients deemed at lower risk for disability who start on first-line MS therapies but experience breakthrough disease, those who switch to a higher-efficacy versus a new first-line therapy have different intermediate-term risk of disability.

DETAILED DESCRIPTION:
FDA-approved multiple sclerosis (MS) disease-modifying therapies (DMTs) target the relapsing phase of MS but have minimal impact once the progressive phase has begun. It is unclear if, in the relapsing phase, there is an advantage of early aggressive therapy with respect to preventing long-term disability. The infectious risks and other complications associated with higher-efficacy treatments highlight the need to quantify their effectiveness in preventing disability.

The TRaditional versus Early Aggressive Therapy for MS (TREAT-MS) trial is a pragmatic, randomized controlled trial that has two primary aims: 1) to evaluate, jointly and independently among patients deemed at higher risk vs. lower risk for disability accumulation, whether an "early aggressive" therapy approach, versus starting with a traditional, first-line therapy, influences the intermediate-term risk of disability, and 2) to evaluate if, among patients deemed at lower risk for disability who start on first-line MS therapies but experience breakthrough disease, those who switch to a higher-efficacy versus a new first-line therapy have different intermediate-term risk of disability.

Hypotheses/Objectives: The main hypothesis is that intermediate-term disability will be reduced by earlier use of higher-efficacy medications. Additional objectives include a) evaluating the magnitude of the treatment effect in patients deemed to be at higher risk versus lower risk of longer-term disability (we hypothesize that the effect size will be greater in the former group) and b) evaluating if, among those without indications of a high risk of longer-term disability, breakthrough disease can be successfully managed by switching to a different first-line therapy or if escalation is required at that time (we hypothesize that switching to a higher-efficacy therapy will be more effective in preventing disability in this group).

There is a great unmet need to identify the most appropriate treatment strategy for people with MS, especially early in the disease course when it may be possible to maximize an individual's chance for preventing long-term disability. There is a paucity of evidence-based guidelines to help clinicians, patients, and payers determine which treatment strategy is best for an individual with MS. Making treatment decisions is a daunting task, and the individualized benefit-risk assessment becomes increasingly difficult as new therapies emerge. Without the availability of direct comparative trials, clinicians and patients are forced to scrutinize observational studies that only provide basic insights into what may be the best treatment path moving forward. It is equally challenging to define what constitutes a suboptimal response to a DMT for an individual patient. Clinicians lack guidance on when to switch therapies and whether to consider a different first-line or if clinicians should escalate immediately to higher-efficacy therapies, so further consensus is needed to determine the optimal time to switch therapies and escalate therapy if an individual is on a first-line therapy from the start. The TREAT-MS trial will help inform patients and the broader health care community on whether patients would most benefit from early, possibly more risky aggressive therapy or if starting with a less aggressive (and, often, less risky) therapy, followed by a switch if breakthrough disease occurs, is warranted. In addition, this study may help identify specific patient populations and/or short-term clinical and paraclinical biomarkers that are strongly predictive of long-term disability that can ensue from MS.

Accrual of sustained disability is the most feared complication for people with MS, and the patient's own perception of their well-being or ill-being has a profound impact on their quality of life. The heterogeneity and unpredictability of MS, along with lack of agreed upon treatment guidelines, augments this fear, leading to a significant negative impact on quality of life. Even patients who are deemed to have "mild" MS experience a significant negative impact on their health-related quality of life that is similar in magnitude to what patients with other severe chronic conditions (i.e., congestive heart failure and chronic obstructive pulmonary disease) report. An extremely important goal for any intervention is to help improve or maintain a high quality of life; therefore, in addition to classic clinical endpoints (e.g. slowing disability progression), the TREAT-MS trial will capture several important and meaningful PROs that will shed light on what treatment strategies may be the best from a patient-centered perspective.

COVID-19 Related Substudy:

Since early 2020, the coronavirus disease 2019 (COVID-19) pandemic has caused clinical care and research disruptions nationwide, including for patients enrolled in the TREAT-MS trial. Many patients with MS, as well as their clinicians, are fearful that MS or the MS therapy they are using may increase the risk or severity of COVID-19 infection. Whether a person with early MS is more likely to experience more severe COVID-19 if treated with a higher-efficacy therapy is not known. Further, whether COVID-19-induced disruptions in therapy or other clinical care increase MS disease activity or MS symptoms is not clear but is relevant, particularly since greater MS activity in the early therapeutic course is associated in observational studies with worse long-term outcomes. Moreover, it is unclear if pre-pandemic anxiety and depression, common comorbidities in people with MS, contribute to decisions to delay care, overall or differently depending on therapeutic strategy (higher-efficacy vs. traditional). TREAT-MS provides an optimal cohort in which to investigate the effect of the COVID-19 pandemic on MS outcomes.

COVID-19 Substudy Aim 1. To evaluate if patients enrolled in TREAT-MS delayed or altered their disease-modifying therapy schedule or other MS care, and whether such alterations are associated with a greater degree of breakthrough inflammatory disease activity or the development of new (or worsening baseline) MS symptoms.

COVID-19 Substudy Aim 2: To evaluate if patients with MS treated with higher-efficacy, versus traditional, therapies differ in the risk of severe COVID-19 infection, defined as requiring hospitalization (with or without intubation) or mortality due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years
* Meets 2017 McDonald criteria for relapsing-remitting MS [patients with clinically isolated syndrome (CIS) are not eligible]
* Must be EITHER John Cunningham (JC) virus antibody negative or low positive (index antibody titer <0.9), OR negative for: Hepatitis B and C, tuberculosis
* HIV negative
* No chemotherapy in past year; if patient has prior history of chemotherapy or malignancy, documentation in chart explaining why potential risks of higher-efficacy therapy are justified

Exclusion Criteria:

* Prior treatment with rituximab, ocrelizumab, ofatumumab, alemtuzumab, mitoxantrone or cladribine
* Prior treatment with any other MS DMT for more than 6 months
* Prior treatment with experimental aggressive therapies (e.g., T-cell vaccine, total lymphoid radiation, stem cells)
* Treatment with teriflunomide within past 2 years (even for ≤ 6 months), unless rapid wash out done (i.e., with cholestyramine or activated charcoal)
* Treatment in the past 6 months with any MS DMT
* Prior treatment with any other investigational immune-modulating /suppressing drug for MS not listed above
* Pregnant or breast-feeding
* Women of child-bearing age who are planning or strongly considering conception during the study time frame

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Time to sustained disability progression | From date of randomization until the date of first documented sustained disability progression, up to 99 months
  Time to sustained disability progression is measured by the Expanded Disability Status Scale plus (EDSS+): a composite endpoint that includes EDSS change (change at any 6 month time point of > or = 1.0 point if baseline EDSS is < or = 5.5 or of > or = 0.5 if baseline EDSS is > or = 6.0, that is sustained 6 months later) OR 20% worsening on either of two specific components of the Multiple Sclerosis Functional Composite (MSFC), the timed 25-foot walk test (T25FWT) and the nine hole peg test (9HPT) that is sustained 6 months later.
Change in Overall Burden of MS | up to 48 weeks from enrollment into COVID-19 related substudy
  The change in overall burden of MS will be defined for the COVID-19 related substudy as the occurrence of breakthrough disease (relapses or new MRI activity) or the development of new (or worsening baseline) MS symptoms, which are (for TREAT-MS) and will continue to be (during the substudy) documented at clinical visits, whether in-person or on tele-visits.

SECONDARY OUTCOMES:
Patient-Determined Disease Steps (PDDS) | up to 99 months
  PDDS is a self-assessment scale of disability due to MS on a scale from 0 to 8 and will be administered as an electronic patient-reported outcome (PRO).
Multiple Sclerosis Functional Composite (MSFC) Composite Score | up to 99 months
  The MSFC consists of the timed 25 foot walk test, the 9-hole peg test, and the Paced Auditory Serial Addition Test (PASAT) and a composite MSFC z-score will be evaluated.
Timed 25 Foot Walk Test | up to 99 months
  Time taken to complete the timed 25 foot walk test, measured twice in units of seconds, will be averaged and evaluated.
Nine-hole Peg Test | up to 99 months
  Time taken to complete the nine-hole peg test, measured twice for each hand (dominant and non-dominant) in units of seconds, will be averaged for each hand and evaluated.
Paced Auditory Serial Addition Test (PASAT) | up to 99 months
  The paced auditory serial addition test that measures processing speed will be administered once; number and percent correct will be evaluated.
Low contrast visual acuity | up to 99 months
  Low-contrast letter acuity (binocular, 2.5% contrast Sloan charts)
Patient-reported incomplete relapse recovery | up to 99 months
  Among participants identified to have a relapse, relapse recovery will be defined as complete or incomplete based on patient self-report.
Neurologic exam-based incomplete relapse recovery | up to 99 months
  Among participants identified to have a relapse, relapse recovery will be defined as complete or incomplete based on neurologic examination (those who have increased Functional System scores, corresponding to the relapse symptoms, of 1.0 point or greater for at least 6 months after the relapse onset, without subsequent accrual of worsening in that same Functional System (e.g. more indicative of progression), will be considered to have incomplete relapse recovery).
Cognition using Symbol Digit Modality Test (SDMT) | up to 99 months
  The SDMT is commonly used in MS to assess processing speed and will be administered orally and used to evaluate changes in cognition throughout the study.
Multiple Sclerosis Impact Scale (MSIS-29) | up to 99 months
  The MSIS-29 will be used to evaluate the impact of MS on the participants and will be administered as an electronic PRO.Multiple Sclerosis Impact Scale (MSIS-29) is an instrument used for measuring the physical (20 items) and psychological (nine items) impact of multiple sclerosis.
Quality of Life in Neurological Disorders (Neuro-QoL): Anxiety Subscale | up to 99 months
  The Anxiety Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Depression Subscale | up to 99 months
  The Depression Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Fatigue Subscale | up to 99 months
  The Fatigue Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Upper Extremity Function | up to 99 months
  The Upper Extremity Function Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Lower Extremity Function | up to 99 months
  The Lower Extremity Function Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Cognitive Function | up to 99 months
  The Cognitive Function Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Positive Affect/Well-being | up to 99 months
  The Positive Affect/Well-being Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Sleep Disturbance | up to 99 months
  The Sleep Disturbance Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Ability to Participate in Social Roles and Activities | up to 99 months
  The Ability to Participate in Social Roles and Activities Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Satisfaction with Social Roles and Activities | up to 99 months
  The Satisfaction with Social Roles and Activities Subscale of Neuro-QoL will be administered as an electronic PRO.
Quality of Life in Neurological Disorders (Neuro-QoL): Stigma | up to 99 months
  The Stigma Subscale of Neuro-QoL will be administered as an electronic PRO.
Employment status | up to 99 months
  The incidence of change in employment to "disabled" or "looking for work, unemployed," will be evaluated for all participants through an electronic PRO.
Marital status | up to 99 months
  Incident divorce or separation, among those who previously were married or in a domestic partnership, will be evaluated for all participants through an electronic PRO.
Serious Adverse Events (SAEs) | up to 99 months
  SAEs (clinically significant infections, malignancies, or the development of other serious comorbidities, as well as unplanned hospitalizations [for non-elective issues, excluding MS relapse] and death)
Adverse event resulting in a decision to change disease-modifying therapy | up to 99 months
  Adverse events meaningful enough to lead to medication discontinuation
Severe COVID-19 Infection | up to 48 weeks from enrollment into COVID-19 related substudy
  Severe COVID-19 infection will be defined as an outcome of "hospitalization or death" due to confirmed or suspected COVID-19 infection

OTHER OUTCOMES:
Brain Magnetic Resonance Imaging (MRI) evidence of neurodegeneration | From 6 months after starting 1st therapy up to 99 months after randomization
  Changes in brain MRI measures of neurodegeneration, including whole brain and normalized gray matter volumes, cortical thickness, subcortical gray matter compartment volumes, and measures of T2 lesion burden.
Number of relapses | up to 99 months
  The number of relapses (new or worsening neurologic symptoms lasting for 24 hours or more in the absence of fever).
Number of new brain lesions on MRI | up to 99 months
  The number of new/enlarging T2-weighted hyperintense lesions and T1-weighted hypointense lesions will be quantified on each MRI scan
Retinal layer thickness by Optical Coherence Tomography (OCT) | up to 99 months
  Retinal nerve fiber layer and ganglion cell/inner plexiform thickness will be evaluated among patients at centers and offices with access to OCT as standard of care
Number of new medications, escalated dosage of medications, and non-pharmacologic interventions for MS-related symptoms | up to 99 months
  As an exploratory outcome, the number of newly-prescribed or dose-escalated medications used for treating MS symptoms (including pain, weakness, numbness/tingling, trouble walking, cognitive problems, fatigue, depression, anxiety, visual dysfunction, spasticity, vertigo, or bladder/bowel/sexual dysfunction) during the trial will be evaluated using the electronic health record. In addition, non-pharmacologic interventions (and referrals to other healthcare providers) for symptom management will also be captured.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M. Mowry, MD, MCR, Principal Investigator — Johns Hopkins University; Scott D. Newsome, DO, Principal Investigator — Johns Hopkins University
Locations (47):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The University of South Alabama, Mobile, Alabama
  - St. Joseph's Hospital & Medical Center - Barrow Neurological Institute, Phoenix, Arizona
  - CommonSpirit Health Research Institute, Carmichael, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida Health, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - The University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - Norton Neurology MS Services, Louisville, Kentucky
  - University of Maryland, Baltimore, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Billings Clinic, Billings, Montana
  - Advanced Neurology Specialists, Great Falls, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York University School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Providence Health and Services - Oregon, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - Vanderbilt Comprehensive MS Center, Nashville, Tennessee
  - Baylor Scott and White Health, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - University of Utah, Salt Lake City, Utah
  - The University of Vermont and State Agricultural College, Burlington, Vermont
  - Blacksburg Neurology, Christiansburg, Virginia
  - Neurology Consultants of Tidewater, Norfolk, Virginia
  - Swedish Health Services, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Kwon S, Sillau S, Corboy JR, Nair KV, Carlson AM. Shifting patterns of multiple sclerosis treatment in a highly prevalent United States population. Ann Clin Transl Neurol. 2024 Jun;11(6):1526-1534. doi: 10.1002/acn3.52069. Epub 2024 Apr 23. PMID 38654416